CLINICAL TRIAL: NCT00726037
Title: A Pilot Study Evaluating the Efficacy of Regulatory T-cell (T-reg) Suppression by Denileukin Diftitox (Ontak) in Metastatic Pancreatic Cancer
Brief Title: A Pilot Study, Evaluating the Efficacy of Regulatory T-cell Suppression by Ontak in Metastatic Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Collaborator withdrew support due to a drug supply interruption.
Sponsor: Loyola University (Other)
Collaborators: Riveria Country Club Organization (Unknown); Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200732
Record Dates: First submitted 2008-07-29; First posted 2008-07-31 (Estimated); Results first posted 2016-08-24 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-08

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: Denileukin diftitox; Metastatic Pancreatic Cancer; Ontak; Regulatory T-cell
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — denileukin diftitox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Three doses of Ontak 9 mcg/Kg IV over 30 minutes every other day for 1 week
  Interventions: Drug: Ontak

INTERVENTIONS:
Drug: Ontak — One dose of Ontak 9 mcg/Kg IV over 30 minutes times 3 doses. 1 dose every other day
  Other Names: Denileukin diftitox

SUMMARY:
This study is designed to determine the duration of T reg suppression in patients with metastatic pancreatic cancer receiving Ontak. The goal is to define the optimal time for future dendritic cell vaccine administration.

DETAILED DESCRIPTION:
Despite improved insight into the epidemiology and biology, pancreatic cancer remains a significant health problem as evidenced by the disappointing survival rates associated with advanced disease. Because of its aggressive growth and early metastatic dissemination, only 20% of patients can be treated by surgery at the time of diagnosis. Furthermore, the overall 5-year survival rate of stage IV disease is < 5% [1-3] despite chemotherapy. With such a dismal outlook, it is obvious that novel treatment strategies are required.

There is limited experience in the literature with the use of Ontak in the treatment of metastatic pancreatic cancer. Viehl, et al, demonstrated in a murine model of pancreatic cancer, that ontak combined with whole tumor vaccine led to a significantly increased T cell-dependent antitumor immune response, as well as an improved survival compared to controls. Our group has an active trial at Loyola evaluating the role of dendritic cell vaccine in patients with unresectable, not metastatic, pancreatic cancer. Preliminary data suggests a correlation with time to progression and restoration of Tregs following an initial decrease after the DC injection. The goal of the current proposal is to determine the time point at which the Tregs reach the nadir within four weeks of ontak injection. When this is determined, we will eventually propose administering ontak followed by DC vaccine at the nadir Treg time point for patients with unresectable pancreatic cancer

ELIGIBILITY:
Inclusion Criteria:

* Male patients and nonpregnant, nonlactating female patient > 18 years old
* Histologic diagnosis of pancreatic cancer with distant disease seen on CT or MRI with no prior chemotherapy or radiotherapy for a least 4 weeks
* Karnofsky performance status equal to or greater than 70%
* Life expectancy of at least 3 months.
* No uncontrolled pain
* No symptoms of bowel obstruction
* Women with child bearing potential must agree to use adequate contraceptives. If she should become pregnant she needs to inform the treating physician
* Ability to give informed consent

Exclusion Criteria:

* Positive serologic testing for HIV, AIDS, human T-cell lymphotrophic virus type 1, hepatitis B, or hepatitis C.
* Hemoglobin <9g/dL; hematocrit <27%; platelets <100,000/ U/L without transfusion support
* Creatinine > 1.8 mg/dL
* Serum albumin < 2.0 mg/dL
* AST > 3X ULN; ALT > 3X ULN
* Bilirubin > 1.8
* Uncontrolled angina, arrhythmias, bronchospasm, hypertension, or hypercalcemia.
* Corticosteroid use within 28 days
* Chemotherapy or radiation within 28 days
* Bacteremia or other signs of active systemic infection
* History of autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margo Shoup, MD, Principal Investigator — Loyola University
Locations (1):
- Loyola Univeristy Medical Center, Cardinal Bernardin Cancer Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Conlon KC, Klimstra DS, Brennan MF. Long-term survival after curative resection for pancreatic ductal adenocarcinoma. Clinicopathologic analysis of 5-year survivors. Ann Surg. 1996 Mar;223(3):273-9. doi: 10.1097/00000658-199603000-00007. PMID 8604907
- [Background] Sperti C, Pasquali C, Piccoli A, Pedrazzoli S. Survival after resection for ductal adenocarcinoma of the pancreas. Br J Surg. 1996 May;83(5):625-31. doi: 10.1002/bjs.1800830512. PMID 8689203
- [Background] Warshaw AL, Fernandez-del Castillo C. Pancreatic carcinoma. N Engl J Med. 1992 Feb 13;326(7):455-65. doi: 10.1056/NEJM199202133260706. No abstract available. PMID 1732772
- [Background] Zwar TD, van Driel IR, Gleeson PA. Guarding the immune system: suppression of autoimmunity by CD4+CD25+ immunoregulatory T cells. Immunol Cell Biol. 2006 Dec;84(6):487-501. doi: 10.1111/j.1440-1711.2006.01471.x. Epub 2006 Sep 5. PMID 16956386
- [Background] Knutson KL, Disis ML, Salazar LG. CD4 regulatory T cells in human cancer pathogenesis. Cancer Immunol Immunother. 2007 Mar;56(3):271-85. doi: 10.1007/s00262-006-0194-y. Epub 2006 Jul 4. PMID 16819631
- [Background] Curiel TJ, Coukos G, Zou L, Alvarez X, Cheng P, Mottram P, Evdemon-Hogan M, Conejo-Garcia JR, Zhang L, Burow M, Zhu Y, Wei S, Kryczek I, Daniel B, Gordon A, Myers L, Lackner A, Disis ML, Knutson KL, Chen L, Zou W. Specific recruitment of regulatory T cells in ovarian carcinoma fosters immune privilege and predicts reduced survival. Nat Med. 2004 Sep;10(9):942-9. doi: 10.1038/nm1093. Epub 2004 Aug 22. PMID 15322536
- [Background] Woo EY, Yeh H, Chu CS, Schlienger K, Carroll RG, Riley JL, Kaiser LR, June CH. Cutting edge: Regulatory T cells from lung cancer patients directly inhibit autologous T cell proliferation. J Immunol. 2002 May 1;168(9):4272-6. doi: 10.4049/jimmunol.168.9.4272. PMID 11970966
- [Background] Griffiths RW, Elkord E, Gilham DE, Ramani V, Clarke N, Stern PL, Hawkins RE. Frequency of regulatory T cells in renal cell carcinoma patients and investigation of correlation with survival. Cancer Immunol Immunother. 2007 Nov;56(11):1743-53. doi: 10.1007/s00262-007-0318-z. Epub 2007 May 9. PMID 17487490
- [Background] Dietl J, Engel JB, Wischhusen J. The role of regulatory T cells in ovarian cancer. Int J Gynecol Cancer. 2007 Jul-Aug;17(4):764-70. doi: 10.1111/j.1525-1438.2006.00861.x. Epub 2007 Feb 16. PMID 17309663
- [Background] Linehan DC, Goedegebuure PS. CD25+ CD4+ regulatory T-cells in cancer. Immunol Res. 2005;32(1-3):155-68. doi: 10.1385/IR:32:1-3:155. PMID 16106066
- [Background] Viehl CT, Moore TT, Liyanage UK, Frey DM, Ehlers JP, Eberlein TJ, Goedegebuure PS, Linehan DC. Depletion of CD4+CD25+ regulatory T cells promotes a tumor-specific immune response in pancreas cancer-bearing mice. Ann Surg Oncol. 2006 Sep;13(9):1252-8. doi: 10.1245/s10434-006-9015-y. Epub 2006 Sep 3. PMID 16952047
- [Background] Ikemoto T, Yamaguchi T, Morine Y, Imura S, Soejima Y, Fujii M, Maekawa Y, Yasutomo K, Shimada M. Clinical roles of increased populations of Foxp3+CD4+ T cells in peripheral blood from advanced pancreatic cancer patients. Pancreas. 2006 Nov;33(4):386-90. doi: 10.1097/01.mpa.0000240275.68279.13. PMID 17079944
- [Background] Hiraoka N, Onozato K, Kosuge T, Hirohashi S. Prevalence of FOXP3+ regulatory T cells increases during the progression of pancreatic ductal adenocarcinoma and its premalignant lesions. Clin Cancer Res. 2006 Sep 15;12(18):5423-34. doi: 10.1158/1078-0432.CCR-06-0369. PMID 17000676
- [Background] Figgitt DP, Lamb HM, Goa KL. Denileukin diftitox. Am J Clin Dermatol. 2000 Jan-Feb;1(1):67-72; discussion 73. doi: 10.2165/00128071-200001010-00008. PMID 11702307
- [Background] Dannull J, Su Z, Rizzieri D, Yang BK, Coleman D, Yancey D, Zhang A, Dahm P, Chao N, Gilboa E, Vieweg J. Enhancement of vaccine-mediated antitumor immunity in cancer patients after depletion of regulatory T cells. J Clin Invest. 2005 Dec;115(12):3623-33. doi: 10.1172/JCI25947. Epub 2005 Nov 23. PMID 16308572

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for this study began on 06/18/2008 and ended on 01/09/2012
Groups:
- Ontak: Three doses of Ontak 9 mcg/Kg IV over 30 minutes every other day for 1 week
Period: Overall Study
Arm/Group | Ontak
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ontak
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: T-reg Suppression From a Fractionated Dose of Ontak in Patients With Metastatic Pancreatic Cancer
Description: The duration of T reg suppression from a fractionated dose of Ontak in patients will be measured in patients with metastatic pancreatic cancer.
Time Frame: days 8, 12 ,19,26 and 33 post administration
Population: Zero participants were analyzed, because the manufacturer withdrew support for the study due to a drug supply interruption
Arm/Group | Ontak
Number analyzed (Participants) | 0

2. Secondary Outcome: Optimal Time for Future Dendritic Cell Vaccine Administration
Description: The goal is to define the optimal time with 95% sensitivity and 95% specificity for future dendritic cell vaccine administration
Time Frame: 33 Days
Population: as for outcome 1
Arm/Group | Ontak
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: For each participant, adverse events were assessed from baseline through end of study (i.e., 33 days)
Arm/Group | Ontak
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

LIMITATIONS AND CAVEATS:
This study was prematurely terminated, because the study drug Ontak is no longer supplied by the manufacturer for this study. Data is not analyzed for any outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No